CLINICAL TRIAL: NCT01408966
Title: Effects of Dark vs. White Chocolate on the Postprandial Increase in Portal Pressure in Cirrhosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Responsible Party: Jaime Bosch /Professor of Medicine, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DarkChocolateinHTP2008
Record Dates: First submitted 2011-08-02; First posted 2011-08-03 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Cirrhosis; Portal Hypertension
Keywords: Dark chocolate; Catechins; Intrahepatic endothelial dysfunction; Cirrhosis; Portal Hypertension
MeSH Terms: conditions — Fibrosis; Hypertension, Portal | interventions — Chocolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DarkChocolate (Experimental): 11 patients were randomized to receiving dark chocolate 0.55 g/kg of body weight (Lindt Excellence 85% Cocoa, Lindt & Sprüngli España) together with the test meal
  Interventions: Dietary Supplement: DarkChocolate
- White chocolate supplementation (Placebo Comparator): 11 patients received 0.63 g/kg white chocolate (Lindt Excellence Natural Vanilla, Lindt & Sprüngli España) in an iso-caloric and iso-volumetric proportion adjusted to body weight.
  Interventions: Dietary Supplement: WhiteChocolate

INTERVENTIONS:
Dietary Supplement: DarkChocolate — Dark chocolatee 0.55 g/kg of body weight was given together with the test meal in sitting position after the baseline measurement of HVPG. The meal + chocolate was ingested in 8 minutes.
  Other Names: Lindt Excellence 85% Cocoa, Lindt & Sprüngli España
  Arms: DarkChocolate
Dietary Supplement: WhiteChocolate — White chocolate 0.63 g/kg white chocolate (Lindt Excellence Natural Vanilla, Lindt & Sprüngli España) in an iso-caloric and iso-volumetric proportion adjusted to body weight was used as a control
  Arms: White chocolate supplementation

SUMMARY:
This study was aimed at testing the hypothesis that supplementing a meal with dark chocolate, which holds potent antioxidant properties, might attenuate the postprandial increase in the hepatic venous pressure gradient (HVPG, clinical equivalent of portal pressure) in patients with cirrhosis

DETAILED DESCRIPTION:
Previous studies showed that the intrahepatic circulation in cirrhosis is not able to adapt to sudden increases in blood flow, such as that occurring after a meal, due to endothelial dysfunction. This leads to a brisk increase in portal pressure (estimated by the HVPG). This method is therefore useful to assess the efficacy of compounds potentially ameliorating intrahepatic endothelial dysfunction. Dark chocolate, which contains a high proportion of cocoa flavonoids such as cathechin and epicatechin- powerful antioxidants, increases NO availability in the systemic circulation and improves systemic endothelial function. We hypothesised that the antioxidant properties of dark chocolate could be beneficial in patients with cirrhosis, since they might improve intrahepatic endothelial dysfunction. Consequently, the aim of this study was to evaluate whether a dark chocolate-containing test meal may attenuate the post-prandial increase in HVPG in patients with cirrhosis and portal hypertension.

HVPG was measured at baseline and 30 minutes after the administration of a test meal supplemented by either dark or white chocolate. Portal vein blood flow and hepatic artery blood flow were measured by Doppler ultrasound. Catechins and NOx were determined for both timepoints.

ELIGIBILITY:
Inclusion Criteria:

1. age over 18 years
2. diagnosis of cirrhosis (proven by biopsy or clinical, laboratory and imaging procedures)
3. presence of esophageal varices of any grade
4. HVPG ≥ 10 mmHg during the hemodynamic study

Exclusion Criteria:

1. food allergy to chocolate
2. ongoing treatment with ascorbic acid and/or other antioxidants
3. diffuse or multinodular hepatocellular carcinoma
4. pregnancy
5. advanced hepatic failure (defined as prothrombin ratio < 40% and bilirubin > 5 mg/dL)
6. renal failure (defined by a serum creatinine level > 1.5 mg/dL)
7. portal vein thrombosis
8. cardiac or respiratory failure
9. previous surgical or transjugular intrahepatic portosystemic shunt

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-08; Primary Completion 2008-10 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Postprandial change in HVPG (% change and absolute change in mmHg) | 30 minutes

SECONDARY OUTCOMES:
Post-prandial change in portal vein blood flow by US-Doppler | 30 minutes
Post-prandial change in nitric oxide metabolites | 30 minutes
Post-prandial changes in catechin and epicatechin | 30 minutes
Post-prandial changes in mean arterial pressure | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Hepatic Hemodynamic Laboratory. Liver Unit. Hospital Clinic., Barcelona, Spain

REFERENCES:
- [Derived] De Gottardi A, Berzigotti A, Seijo S, D'Amico M, Thormann W, Abraldes JG, Garcia-Pagan JC, Bosch J. Postprandial effects of dark chocolate on portal hypertension in patients with cirrhosis: results of a phase 2, double-blind, randomized controlled trial. Am J Clin Nutr. 2012 Sep;96(3):584-90. doi: 10.3945/ajcn.112.040469. Epub 2012 Jul 18. PMID 22811444